CLINICAL TRIAL: NCT05842057
Title: Phase 2 Randomized Trial: Human Amnion Membrane Allograft and Early Return of Erectile Function After Radical Prostatectomy (HAMMER)
Brief Title: Human Amnion Membrane Allograft and Early Return of Erectile Function After Radical Prostatectomy
Acronym: HAMMER
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Integra LifeSciences Corporation (Industry)
Responsible Party: Principal Investigator, Sanoj Punnen, MD, MAS, Associate Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20220852
Record Dates: First submitted 2023-04-24; First posted 2023-05-03 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer; Erectile Dysfunction Following Radical Prostatectomy
Keywords: Prostatectomy; Allograft Membrane
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants will be blinded to the treatment they receive. To minimize bias on the surgical team during the nerve sparing process, the surgical team will be blinded to arm allocation until after the prostate is removed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Membrane Arm: dHACM Group (Experimental): Participants will undergo standard of care robot-assisted radical prostatectomy (RARP) surgery and the dehydrated Human Amnion Chorion Membrane (dHACM) membrane placed after removal of the prostate. Participants will be in the group for approximately 12 months.
  Interventions: Biological: BioDFence G3 Placental Tissue Membrane; Procedure: Robot-Assisted Radical Prostatectomy
- Control Arm: No dHACM Group (Other): Participants will undergo standard of care RARP surgery but will have no dehydrated Human Amnion Chorion Membrane (dHACM) placed after removal of the prostate. Participants will be in the group for approximately 12 months.
  Interventions: Procedure: Robot-Assisted Radical Prostatectomy

INTERVENTIONS:
Biological: BioDFence G3 Placental Tissue Membrane — The BioDFence G3 Placental Tissue Membrane is a three-layer tissue allograft consisting of amnion-chorion-amnion. Amniotic membranes will be placed over the neurovascular bundle after extirpative RARP. The membrane will be cut into two longitudinal pieces and placed over each neurovascular bundle separately.
  Other Names: Dehydrated Human Amnion Chorion Membrane (dHACM); Human Amnion Membrane Allograft
  Arms: Membrane Arm: dHACM Group
Procedure: Robot-Assisted Radical Prostatectomy — Robot-assisted surgical removal of the prostate, administered standard of care.
  Other Names: RARP

SUMMARY:
The purpose of this research study is to evaluate if placing a dehydrated human amnion chorion membrane (dHACM) over the nerves after removal of the prostate during surgery (radical prostatectomy) will allow an earlier recovery of erectile function and urinary control after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 40 to 80 years with localized prostate cancer who are undergoing RARP at the University of Miami (UM).

Exclusion Criteria:

1. Men requiring the use of any non-oral erectile aids for erectile dysfunction (ED).
2. Men with baseline EPIC26 scores < 50.
3. Patients with complete, bilateral nerve resection.
4. Previous treatment for prostate cancer.
5. Previous history of pelvic radiation.
6. Patients with impaired decision-making capacity.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Erectile Function Recovery as Measured by EPIC26 Sexual Domain Score | Baseline, 12 Months Post-RARP
  Erectile function recovery among participants will be measured by the change in scores within the Sexual Domain of the Expanded Prostate Cancer Index Composite Short Form (EPIC26). The EPIC26 is a 26-item questionnaire used to measure health-related quality of life (HRQOL) among men with prostate cancer. The EPIC26 has five domains: Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal. Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale with higher scores representing better HRQOL.

SECONDARY OUTCOMES:
Change in Erectile Function Recovery as Measured by SHIM Score | Baseline, 12 Months Post-RARP
  Erectile function recovery among participants will be measured as the change in Sexual History Inventory for Men (SHIM). The SHIM is a health-related quality of life (HRQOL) questionnaire whose scores measure the severity of erectile dysfunction (ED) in men using points on a scale. The minimum score of 1 to 7 points indicates severe ED; a score of 8 to 11 points indicates moderate ED; a score of 12 to 15 points indicates mild-to-moderate ED; a score of 17 to 21 points indicates mild ED; and the maximum score of 22 to 25 points indicates no significant ED.
Change in Proportion of Men with Mild ED or Better as Defined by EPIC26 Sexual Domain Score | Baseline, 3 months, 6 months, 9 months, 12 months Post-RARP
  Proportion of men with mild ED or better as defined by an EPIC26 Sexual Domain score greater than or equal to 60. Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale with higher scores representing better sexual function.
Change in Proportion of Participants with mild ED or Better as Defined by SHIM Score | Baseline, 3 months, 6 months, 9 months, 12 months Post-RARP
  Proportion of participants with mild ED or better as defined by a SHIM score greater than or equal to 17. The SHIM is a health-related quality of life (HRQOL) questionnaire whose scores measure the severity of erectile dysfunction (ED) in men using points on a scale. The minimum score of 1 to 7 points indicates severe ED; a score of 8 to 11 points indicates moderate ED; a score of 12 to 15 points indicates mild-to-moderate ED; a score of 17 to 21 points indicates mild ED; and the maximum score of 22 to 25 points indicates no significant ED.
Change in Proportion of Participants with Erections Adequate for Penetration ≥ 50% of the time | Baseline, 3 months, 6 months, 9 months, 12 months Post-RARP
  Proportion of participants with erections adequate for penetration greater than or equal to 50-percent of the time.
Change in Proportion of Participants who Require the Use of More Invasive Erectile Aids | Baseline, 3 months, 6 months, 9 months, 12 months Post-RARP
  Proportion of participants who require the use of more invasive erectile aids (intra-cavernosal injection, vacuum pump, or penile prosthesis).
Change in Rate of Urinary Control | Baseline, 3 months, 6 months, 9 months, 12 months Post-RARP
  Rate of urinary control as measured by EPIC26 question 3 that reports the number of participants requiring no pads per day.
Change in Biochemical Failure | Baseline, 3 months, 6 months, 9 months, 12 months Post-RARP
  Biochemical failure among participants will measured as a prostate-specific antigen (PSA) level > 0.2 ng/ml on two consecutive samples.
Number of Treatment-Related Adverse Events | Up to 12 months post-RARP
  The number of treatment-related adverse events among participants will be assessed by treating physician using the Clavien-Dindo grading scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sanoj Punnen, MD, MAS, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No